CLINICAL TRIAL: NCT01993186
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Study to Assess the Safety and Efficacy of UX007 in Subjects With Glucose Transporter Type 1 Deficiency Syndrome
Brief Title: Phase 2 Study of Triheptanoin (UX007) for the Treatment of Glucose Transporter Type 1 Deficiency Syndrome (Glut1 DS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX007G-CL201
Expanded Access: NCT03773770 (Available)
Record Dates: First submitted 2013-10-31; First posted 2013-11-25 (Estimated); Results first posted 2020-05-29 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome (Glut1 DS)
Keywords: Glucose Transporter Type 1 Deficiency Syndrome Glut1
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UX007 (Experimental): Participants randomized to receive UX007 enter a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
  Following completion of the Week 8 study visit, participants continue treatment with open-label UX007 at the 35% dose level for an additional 44 weeks (Weeks 8-52).
  Interventions: Drug: UX007
- Placebo (Placebo Comparator): Participants randomized to receive placebo enter a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
  Following completion of the Week 8 study visit, placebo participants continue treatment with open-label UX007 at the 35% dose level for an additional 44 weeks (Weeks 8-52).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UX007 — oral liquid
  Other Names: C7 oil; triheptanoin; glycerol triheptanoate; glycerol trienanthate; 1, 2, 3-trienanthoylglycerol; trienanthin; 2,3-di(heptanoyloxy)propyl heptanoate
  Arms: UX007
Drug: Placebo — oral liquid
  Arms: Placebo

SUMMARY:
The primary objectives of the study are to evaluate the efficacy of UX007 compared to placebo as measured by the reduction from randomization to Week 8 in frequency of seizures and to evaluate the safety of UX007 via adverse event (AE) rates, laboratory values, and electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Glut1 DS confirmed by SLC2A1 mutation
2. Males and females at least 1 of age at the time of informed consent
3. Average of at least 2 observable seizures (generalized or partial-onset [simple partial motor, complex partial, absence, or secondarily generalized seizures) in 4 weeks over the last 24 weeks, by subject or caregiver report
4. At least 2 observable seizures (generalized or partial-onset [simple partial motor, complex partial, or secondarily generalized seizures) in 4 weeks during the Baseline Period, with no 3-week seizure-free period during the Baseline Period OR absence seizures documented on Screening electroencephalogram (EEG)
5. Continuing to have seizures despite a prior or current use of at least 1 antiepileptic drug (AED)
6. Allowed to be on up to 3 concomitant AEDs that must have been stable in dose at least 2 weeks prior to the beginning of screening and anticipated to remain stable in dose through the end of the 8-week, placebo-controlled Treatment Period
7. Not on, or not fully compliant with a prescribed diet plan (e.g. KD)
8. Plasma level of beta-hydroxybutyrate (BHB) ≤ 1 mmol/L (non-fasting) at Screening
9. Provide written or verbal assent (if possible) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures
10. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, comply with accurate completion of the seizures diary, and likely to complete the 8 week, placebo-controlled, Treatment Period
11. Females of childbearing potential must have a negative pregnancy test at Screening, be willing to use an acceptable method of contraception, and have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have not reached menarche, had total hysterectomy, have been in menopause for at least two years, or have had tubal ligation at least one year prior to Screening.

Exclusion Criteria:

1. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels exceeding 3 times the upper limit of normal at Screening
2. Any known hypersensitivity to triheptanoin or safflower oil that, in the judgment of the investigator, places the subject at increased risk for adverse effects
3. Prior use of triheptanoin within 30 days prior to Screening
4. History of, or current suicidal ideation, behavior and/or attempts
5. Pregnant and/or breastfeeding an infant at Screening
6. Participants unwilling or unable to discontinue use of a prohibited medication or other substance that may confound study objectives
7. Use of any investigational product (drug or supplement, including medium chain triglyceride [MCT] oil) within 30 days prior to Screening, or at any time during the study
8. Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment
9. Has a concurrent disease or condition, or laboratory abnormality that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduces additional safety concerns (e.g., diabetes mellitus, other concurrent neurological or psychiatric disorders)

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (14):
- United States (8):
  - Children's Hospital Colorado - University of Colorado, Denver, School of Medicine, Aurora, Colorado
  - Miami Children's Research Institute, Miami, Florida
  - Neurology & Epilepsy Research Center, Orlando, Florida
  - Columbia University - Department of Neurology, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cook Children's Hospital, Fort Worth, Texas
  - University of Texas Neurometabolic Clinic, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Melbourne Brain Centre, Heidelberg, Victoria, Australia
- Service de Neurologie Pédiatrique et des Maladies Métaboliques - INSERM U1141 Hôpital Robert Debré - APHP, Paris, Cedex 19, France
- Sheba University Medical Center, Tel Aviv, Israel
- Unita' Operativa Neurologia Pediatrica e Malattie Muscolari Istituto "Giannina Gaslini", Genova, Italy
- Hospital Sant Joan de Deu, Barcelona, Spain
- Newcastle University, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Striano P, Auvin S, Collins A, Horvath R, Scheffer IE, Tzadok M, Miller I, Kay Koenig M, Lacy A, Davis R, Garcia-Cazorla A, Saneto RP, Brandabur M, Blair S, Koutsoukos T, De Vivo D. A randomized, double-blind trial of triheptanoin for drug-resistant epilepsy in glucose transporter 1 deficiency syndrome. Epilepsia. 2022 Jul;63(7):1748-1760. doi: 10.1111/epi.17263. Epub 2022 May 21. PMID 35441706
- See also: Related Info — http://www.ultragenyx.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Beginning with the Screening visit, participants recorded seizure frequency during a 6-week Baseline Period. If the participant did not meet the seizure count criteria, the participant was considered a screen failure and was not randomized.
Groups:
- UX007: Participants randomized to receive UX007 entered a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
  Following completion of the Week 8 study visit, participants continued treatment with open-label UX007 at the 35% dose level for an additional 44 weeks (Weeks 8-52).
- Placebo: Participants randomized to receive placebo entered a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
  Following completion of the Week 8 study visit, placebo participants continued treatment with open-label UX007 at the 35% dose level for an additional 44 weeks (Weeks 8-52).
Period: Double-Blind Placebo-Controlled Period
Arm/Group | UX007 | Placebo
Started | 25 | 11
Completed | 23 | 11
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open-Label Extension Period
Arm/Group | UX007 | Placebo
Started | 23 | 11
Completed | 16 | 5
Not Completed | 7 | 6
Not completed — Other, Not Specified | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Principal Investigator Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Subject Non-Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UX007 | Placebo | Total
Number analyzed (Participants) | 25 | 11 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.86 (5.107) | 15.24 (13.795) | 14.28 (8.525)
Age, Customized [Count of Participants; unit: Participants]
  2 years to < 12 years | 8 | 7 | 15
  12 years to < 18 years | 12 | 1 | 13
  18 years to < 65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 23 | 9 | 32
  Other (Not Specified) | 1 | 0 | 1
Total Seizure Frequency Per 4 Weeks [Median (Full Range); unit: seizures per 4 weeks] — Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. Absence seizures from electroencephalography (EEG) include absence awake (>=10sec), absence sleep (>=10sec), indeterminate absence awake (3-10sec), and indeterminate absence sleep (3-10sec).
  seizures per 4 weeks | 96.6 [0 to 10250] | 2.1 [0 to 1176] | 35.7 [0 to 10250]

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction From Baseline to Week 8 in Frequency of Total Seizures (Normalized to a 4-Week Rate)
Description: Reduction from baseline to Week 8 in frequency of seizures (normalized to a 4-week rate): observable seizures measured for 6 weeks after 2-week titration by diary and absence seizures measured overnight by EEG. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. Absence seizures from EEG include absence awake (>=10 sec), absence sleep (>=10 sec), indeterminate absence awake (3-10 sec), and indeterminate absence sleep (3-10 sec). A negative value indicates an increase in frequency.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product.
Measure: Median (Full Range); unit: percent reduction of seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
percent reduction of seizures per 4 wks | 12.6 [-651 to 100] | 0.0 [-1021 to 100]
Statistical Analysis 1: Comparison: UX007 vs Placebo; Non-parametric post-hoc analysis: Hodges-Lehmann estimate of the location shift with 90% confidence interval (CI) and Wilcoxon Rank Sum test p-value, based on Wilcoxon rank-sum test; Test type: Superiority; p = 0.5812, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 13.45, 90% CI 2-sided [-38.63 to 80.95]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Discontinuations Due to TEAEs During the Placebo-Controlled Period
Description: An adverse event (AE) was defined as any untoward medical occurrence, whether or not considered drug related. A serious AE was defined as an AE or suspected adverse reaction that at any dose resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, or an important medical event that may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed in the definition. An AE was considered a TEAE if it occurred or worsened in severity on or after the date of the first dose of study drug. An AE was considered a UX007 emergent adverse event if it occurred or worsened in severity on or after the first date of first dose of UX007 during the study.
Time Frame: Weeks 0 to 8
Population: Safety Analysis Set: all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
Participants
  TEAE | 22 | 9
  Serious TEAE | 1 | 0
  Grade 3 or 4 TEAE | 2 | 0
  TEAE Leading to Study Discontinuation | 0 | 0
  TEAE Leading to Death | 0 | 0
  Gastrointestinal TEAE | 18 | 5
  Related TEAE | 18 | 5
  Related Serious TEAE | 0 | 0
  Related Gastrointestinal TEAE | 17 | 4
  UX007 Emergent AE | 22 | 0
  Serious UX007 Emergent AE | 1 | 0

3. Primary Outcome: Number of Participants With TEAEs, Serious TEAEs and Discontinuations Due to TEAEs During the Extension Period
Description: An AE was defined as any untoward medical occurrence, whether or not considered drug related. A serious AE was defined as an AE or suspected adverse reaction that at any dose resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, or an important medical event that may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed in the definition. An AE was considered a TEAE if it occurred or worsened in severity on or after the date of the first dose of study drug. An AE was considered a UX007 emergent adverse event if it occurred or worsened in severity on or after the first date of first dose of UX007 during the study.
Time Frame: Weeks 9 to 52 plus 30 days
Population: Safety Analysis Set: all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 23 | 11
Participants
  TEAE | 21 | 11
  Serious TEAE | 2 | 0
  Grade 3 or 4 TEAE | 1 | 0
  TEAE Leading to Study Discontinuation | 1 | 0
  TEAE Leading to Death | 0 | 0
  Gastrointestinal TEAE | 15 | 10
  Related TEAE | 19 | 8
  Related Serious TEAE | 0 | 0
  Related Gastrointestinal TEAE | 13 | 8
  UX007 Emergent AE | 21 | 11
  Serious UX007 Emergent AE | 2 | 0

4. Secondary Outcome: Percent Reduction From Baseline to Week 8 in Frequency of Observable Seizures (Normalized to a 4-Week Rate)
Description: Reduction from baseline to Week 8 in frequency of seizures (normalized to a 4-week rate): observable seizures measured for 6 weeks after 2-week titration by diary. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. A negative value indicates an increase in frequency.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product. Participants with observable seizures.
Measure: Median (Full Range); unit: percent reduction in seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 17 | 10
percent reduction in seizures per 4 wks | 0.0 [-651 to 84] | 0.0 [-1021 to 75]
Statistical Analysis 1: Comparison: UX007 vs Placebo; Non-parametric post-hoc analysis: Hodges-Lehmann estimate of the location shift with 90% CI and Wilcoxon Rank Sum test p-value, based on Wilcoxon rank-sum test; Test type: Superiority; p = 0.8197, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0, 90% CI 2-sided [-51.23 to 84.25]

5. Secondary Outcome: Percent Reduction From Baseline to Week 8 in Frequency of Absence Seizures (Normalized to a 4-Week Rate)
Description: Reduction from baseline to Week 8 in frequency of absence seizures measured overnight by EEG. Absence seizures from EEG include absence awake (>=10 sec), absence sleep (>=10 sec), indeterminate absence awake (3-10 sec), and indeterminate absence sleep (3-10 sec). A negative value indicates an increase in frequency.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product. Participants with absence seizures.
Measure: Median (Full Range); unit: percent reduction in seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 17 | 6
percent reduction in seizures per 4 wks | 0.0 [-2400 to 100] | 0.0 [0 to 100]
Statistical Analysis 1: Comparison: UX007 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7276, Wilcoxon rank-sum test; Hodges-Lehmann estimate = 0, 90% CI 2-sided [0 to 37.5]

6. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline to Week 8 in Frequency of Total Seizures
Description: Seizure response, defined as the percentage of participants with at least 50% reduction from randomization to Week 8 in frequency of total seizures. Includes observable generalized and partial-onset seizures measured for 6 weeks by diary and absence seizures measured overnight by EEG. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. Absence seizures from EEG include absence awake (>=10 sec), absence sleep (>=10 sec), indeterminate absence awake (3-10 sec), and indeterminate absence sleep (3-10 sec).
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
percentage of participants | 20.0 | 36.4

7. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline to Week 8 in Frequency of Observable Seizures
Description: Observable seizure response, defined as the percentage of participants with at least 50% reduction from randomization to Week 8 in frequency of observable seizures. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological.
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 17 | 10
percentage of participants | 5.9 | 30.0

8. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline to Week 8 in Frequency of Absence Seizures
Description: Absence seizure response, defined as the percentage of participants with at least 50% reduction from randomization to Week 8 in frequency of absence seizures. Absence seizures from EEG include absence awake (>=10 sec), absence sleep (>=10 sec), indeterminate absence awake (3-10 sec), and indeterminate absence sleep (3-10 sec).
Time Frame: Baseline, Week 8
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 17 | 6
percentage of participants | 23.5 | 16.7

9. Secondary Outcome: Change From Baseline to Week 8 in Cambridge Neuropsychological Test Automated Battery (CANTAB), Reaction Time (RTI) Scores, Generalized Estimating Equation (GEE)
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. RTI Simple choice reaction time standard deviation (RTISRTSD) assesses the cognitive domain of attention, with scores on a continuous range from 0 to 5000; lower scores indicate better function. RTI median simple choice reaction time (RTIMDSRT) assesses the cognitive domain of reaction time, with scores on a continuous range from 100 to 5100; lower scores indicate better function. RTI median 5-choice reaction time (RTIMDFRT) assesses the cognitive domain of reaction time, with scores on a continuous range from 100 to 5100; lower scores indicate better function. GEE statistical model.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set, CANTAB: Subset of participants taking UX007 during the treatment period in the efficacy analysis set who had a baseline and at least 1 post baseline (Week 4 or Week 8) CANTAB assessment performed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
score on a scale
  RTISRTSD | 41.698 (42.3539) | 44.082 (53.3552)
  RTIMDSRT | 15.512 (15.9204) | -48.157 (48.8781)
  RTIMDFRT | -14.723 (14.1862) | 49.112 (58.4722)
Statistical Analysis 1: Comparison: UX007 vs Placebo; RTISRTSD; Test type: Superiority; p = 0.486, GEE model — One-sided p-value. Additional model covariates include the corresponding baseline CANTAB score, visit and the interaction between visit and treatment; Least squares mean difference = -2.384, 90% CI 2-sided [-114.44 to 109.67], Standard Error of Mean 68.1231
Statistical Analysis 2: Comparison: UX007 vs Placebo; RTIMDSRT; Test type: Superiority; p = 0.8849, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = 63.669, 90% CI 2-sided [-23.6 to 150.94], Standard Error of Mean 53.0537
Statistical Analysis 3: Comparison: UX007 vs Placebo; RTIMDFRT; Test type: Superiority; p = 0.1463, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = -63.835, 90% CI 2-sided [-163.59 to 35.93], Standard Error of Mean 60.6496

10. Secondary Outcome: Change From Baseline to Week 8 in CANTAB, Paired Associates Learning (PAL) Scores, GEE
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. PAL total errors adjusted (PALTEA) assesses the cognitive domain of episodic memory/new learning, with scores on a discrete, ordinal scale from 0 to 137; lower scores indicate better function. PAL first trial memory score (PALFTMS) assesses the cognitive domain of episodic memory, with scores on a discrete, ordinal scale from 0 to 27; higher scores indicate better function. GEE statistical model.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
score on a scale
  PALTEA | -10.082 (2.4784) | -27.849 (11.3061)
  PALFTMS | 2.574 (0.6833) | 3.105 (2.0766)
Statistical Analysis 1: Comparison: UX007 vs Placebo; PALTEA; Test type: Superiority; p = 0.9378, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = 17.768, 90% CI 2-sided [-1.26 to 36.79], Standard Error of Mean 11.5659
Statistical Analysis 2: Comparison: UX007 vs Placebo; PALFTMS; Test type: Superiority; p = 0.5959, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = -0.531, 90% CI 2-sided [-4.13 to 3.06], Standard Error of Mean 2.1853

11. Secondary Outcome: Change From Baseline to Week 8 in CANTAB, Spatial Span (SSP) Span Length Scores, GEE
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. SSP Span Length (SSPSLF) assesses the cognitive domain of sequential memory, with scores on a discrete, ordinal scale from 2 to 9; higher scores indicate better function. GEE statistical model.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
score on a scale | 0.019 (0.2387) | -0.041 (0.4246)
Statistical Analysis 1: Comparison: UX007 vs Placebo; SSPSLF; Test type: Superiority; p = 0.4522, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = 0.06, 90% CI 2-sided [-0.76 to 0.88], Standard Error of Mean 0.4988

12. Secondary Outcome: Change From Baseline to Week 8 in CANTAB, Spatial Working Memory (SWM) Scores, GEE
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. SWM between errors (SWMBE48) assesses the cognitive domain of working memory, with scores on a discrete, ordinal scale from 0 to 360; lower scores indicate better function. SWM strategy (SWMS68) assesses the cognitive domain of executive function/strategy, with scores on a discrete, ordinal scale from 4 to 28; lower scores indicate better function. GEE statistical model.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 25 | 11
score on a scale
  SWMBE48 | 1.003 (1.4582) | 2.240 (1.8036)
  SWMS68 | 0.060 (0.4794) | 0.022 (0.4279)
Statistical Analysis 1: Comparison: UX007 vs Placebo; SWMBE48; Test type: Superiority; p = 0.3017, GEE model — [p-value comment as in outcome 9, analysis 1]; LS Mean Difference = -1.237, 90% CI 2-sided [-5.15 to 2.68], Standard Error of Mean 2.381
Statistical Analysis 2: Comparison: UX007 vs Placebo; SWMS68; Test type: Superiority; p = 0.5235, GEE model — [p-value comment as in outcome 9, analysis 1]; Least squares mean difference = 0.038, 90% CI 2-sided [-1.03 to 1.11], Standard Error of Mean 0.6495

13. Secondary Outcome: Change From Baseline to Week 8 in Distance Traveled (in Meters) as Measured by 6-Minute Walk Test (6MWT)
Description: Participants were instructed to walk the length of a pre-measured 20-30 meter course in a hallway for 6 consecutive minutes. The total distance walked (meters) in a 6 minute period was recorded.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set - 6MWT: Subset of participants taking UX007 during the treatment period in the efficacy analysis set who had a baseline and at least 1 post baseline (Week 4 or Week 8) 6MWT assessment performed.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 23 | 11
meters | -10.336 (14.8614) | -3.439 (16.1506)
Statistical Analysis 1: Comparison: UX007 vs Placebo; 6MWT distance traveled; Test type: Superiority; p = 0.6205, GEE model — One-sided p-value. Additional model covariates include the corresponding baseline value, visit and the interaction between visit and treatment; Least squares mean difference = -6.897, 90% CI 2-sided [-43.874 to 30.08], Standard Error of Mean 22.4806

14. Secondary Outcome: Change From Baseline to Week 8 in Distance Traveled (in Percent Predicted) as Measured by 6MWT
Description: Participants were instructed to walk the length of a pre-measured 20-30 meter course in a hallway for 6 consecutive minutes. The total distance walked (meters) in a 6 minute period was recorded. The percent of predicted normal distance walked was determined based on published normative data.
Time Frame: Baseline, Week 8
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: percent of predicted distance
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 23 | 11
percent of predicted distance | -1.338 (2.4752) | 0.016 (2.6398)
Statistical Analysis 1: Comparison: UX007 vs Placebo; 6MWT distance traveled (percent predicted); Test type: Superiority; p = 0.6476, GEE model — [p-value comment as in outcome 13, analysis 1]; Least squares mean difference = -1.354, 90% CI 2-sided [-7.236 to 4.527], Standard Error of Mean 3.5759

15. Secondary Outcome: Time (in Minutes) to Onset of Paroxysmal Exertional Dyskinesia (PED) as Measured During 6MWT Over Time Through Week 8
Description: For the 6MWT, subjects were instructed to walk the length of a pre-measured 20-30 meter course in a hallway for 6 consecutive minutes. The total distance walked (meters) in a 6 minute period was recorded. PED occurring during the 6MWT was assessed. (PED is characterized by transient abnormal, involuntary movements primarily affecting the legs and feet, and typically precipitated by prolonged exertion.)
Time Frame: Baseline, Week 4, Week 8
Population: Efficacy Analysis Set - 6MWT: Subset of participants taking UX007 during the treatment period in the efficacy analysis set who had a baseline and at least 1 post baseline (Week 4 or Week 8) 6MWT assessment performed. Participants with at least 1 PED.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 3 | 0
minutes
  Week 4 | 4.7 (4.73) |
  Week 8 | 1.8 (1.30) |

16. Secondary Outcome: Change From Baseline to Week 8 in Gross Motor Function Measure-88 (GMFM-88) Total Score
Description: The GMFM-88 is a standardized observational measure of abilities that includes the following 5 domains: lying/rolling, sitting, crawling/kneeling, standing, and walking/running/jumping. The GMFM-88 scores include the following:
  * Lying & Rolling Score, Range 0-100%, higher is better
  * Sitting Score, Range 0-100%, higher is better
  * Crawling & Kneeling Score, Range 0-100%, higher is better
  * Standing Score, Range 0-100%, higher is better
  * Walking, Running & Jumping Score, Range 0-100%, higher is better
  * Total Score = (Sum of 5 Above Scores) / 5, Range 0-100%, higher is better.
Time Frame: Baseline, Week 8
Population: Efficacy Analysis Set - GMFM-88: Subset of participants taking UX007 during the treatment period in the efficacy analysis set who had a baseline and at least 1 post baseline (Week 4 or Week 8) GMFM-88 assessment performed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 21 | 11
score on a scale | 3.209 (2.3669) | 1.642 (2.6690)
Statistical Analysis 1: Comparison: UX007 vs Placebo; GMFM-88 UX007-Placebo; Test type: Superiority; p = 0.3435, GEE model — One-sided p-value. Additional model covariates include baseline GMFM-88 total score, visit and the interaction between visit and treatment; Least squares mean difference = 1.568, 90% CI 2-sided [-4.83 to 7.97], Standard Error of Mean 3.8899

17. Secondary Outcome: Percent Reduction From Baseline Over Time in Frequency of Total Seizures (Normalized to a 4-Week Rate)
Description: Reduction from baseline over time in frequency of seizures (normalized to a 4-week rate): observable seizures measured for 6 weeks after 2-week titration by diary and absence seizures measured overnight by EEG. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. Absence seizures from EEG include absence awake (>=10 sec), absence sleep (>=10 sec), indeterminate absence awake (3-10 sec), and indeterminate absence sleep (3-10 sec). A negative value indicates an increase in frequency.
Time Frame: Baseline, Week 26, Week 31
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product. Participants with an assessment at given time point.
Measure: Median (Full Range); unit: percent reduction of seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 22 | 11
percent reduction of seizures per 4 wks
  Week 26 | 7.8 [-409 to 100] | 0.0 [-207 to 94]
  Week 31: number analyzed (Participants) | 19 | 8
  Week 31 | 42.7 [-267 to 100] | 5.3 [-681 to 75]

18. Secondary Outcome: Percent Reduction From Baseline Over Time in Frequency of Observable Seizures (Normalized to a 4-Week Rate)
Description: Reduction from baseline over time in frequency of seizures (normalized to a 4-week rate): observable seizures measured for 6 weeks after 2-week titration by diary. Observable seizures from the diary include generalized tonic-clonic, generalized tonic, generalized clonic, generalized atonic, partial/focal with secondary generalization, myoclonic, myoclonic (astatic) atonic, myoclonic tonic, complex partial/focal, simple partial/focal motor, simple partial/focal sensory, and simple partial/focal psychological. A negative value indicates an increase in frequency.
Time Frame: Baseline, Week 26, Week 31, Week 36, Week 52
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product. Participants with observable seizures and an assessment at given time point.
Measure: Median (Full Range); unit: percent reduction in seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 15 | 10
percent reduction in seizures per 4 wks
  Week 26 | 0.0 [-260 to 88] | -27.7 [-207 to 74]
  Week 31: number analyzed (Participants) | 12 | 7
  Week 31 | 23.6 [-267 to 100] | 0.0 [-681 to 67]
  Week 36: number analyzed (Participants) | 12 | 7
  Week 36 | 42.5 [-438 to 100] | -49.8 [-400 to 77]
  Week 52: number analyzed (Participants) | 12 | 6
  Week 52 | 31.0 [-222 to 100] | -10.3 [-358 to 85]

19. Secondary Outcome: Percent Reduction From Baseline Over Time in Frequency of Absence Seizures (Normalized to a 4-week Rate)
Description: as for outcome 5
Time Frame: Baseline, Week 26, Week 31
Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational product. Participants with absence seizures and an assessment at given time point.
Measure: Median (Full Range); unit: percent reduction in seizures per 4 wks
Arm/Group | UX007 | Placebo
Number analyzed (Participants) | 14 | 4
percent reduction in seizures per 4 wks
  Week 26 | 0.0 [-3135 to 100] | 0.0 [0 to 94]
  Week 31: number analyzed (Participants) | 12 | 3
  Week 31 | 0.0 [-3905 to 100] | 0.0 [0 to 75]

ADVERSE EVENTS:
Time Frame: Placebo-controlled period from first dose of study drug through Week 8. Extension period: Week 9 up to Week 52 plus 30 days.
Groups:
- Placebo Controlled Period / UX007: Participants randomized to receive UX007 entered a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
- Placebo Controlled Period / Placebo: Participants randomized to receive placebo entered a 2-week dose titration period to achieve study drug treatment comprising up to 35% of total daily calories or to the maximum tolerated dose level and maintained at the 35% total daily calorie dose level for a 6-week treatment period.
- Extension Period / UX007: Following completion of the Week 8 study visit, placebo and UX007 participants continued treatment with open-label UX007 at the 35% dose level for an additional 44 weeks (Weeks 8-52).
Arm/Group | Placebo Controlled Period / UX007 | Placebo Controlled Period / Placebo | Extension Period / UX007
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/11 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/11 | 2/34
Other Adverse Events (participants affected / at risk) | 21/25 | 9/11 | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period / UX007 (N=25) | Placebo Controlled Period / Placebo (N=11) | Extension Period / UX007 (N=34)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period / UX007 (N=25) | Placebo Controlled Period / Placebo (N=11) | Extension Period / UX007 (N=34)
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 0 | 5
Breath Odour (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 3 | 18
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 5 | 0 | 5
Vomiting (Gastrointestinal disorders) | 11 | 2 | 15
Pyrexia (General disorders) | 2 | 0 | 6
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 2
Otitis Media Acute (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1 | 6
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lip Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight Increased (Investigations) | 3 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Clonic Convulsion (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 3
Seizure (Nervous system disorders) | 0 | 0 | 2
Abnormal Behaviour (Psychiatric disorders) | 0 | 0 | 3
Agitation (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT01993186/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT01993186/SAP_001.pdf